CLINICAL TRIAL: NCT03879421
Title: The Role of Anterior Segment Optical Coherence Tomography in Evaluation of the Keratoconic Cornea After Corneal Collagen Cross Linking.
Brief Title: Evaluation of the Keratoconic Cornea After Corneal Collagen Cross Linking.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Reham Mahmoud Abdelrahman (Other)
Responsible Party: Sponsor-Investigator, Reham Mahmoud Abdelrahman, Principal Investigator, Assiut University
Organization: Assiut University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TROASOCTIEOTKCACCCL
Record Dates: First submitted 2019-03-13; First posted 2019-03-18 (Actual); Last update posted 2019-03-19 (Actual); Status verified 2019-03

CONDITIONS: Keratoconus
MeSH Terms: conditions — Keratoconus

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Epithelium-off accelerated CXL) (Active Comparator): patients with corneal thickness > 400 µm (thinnest location) were assigned into Epi-off accelerated CXL procedure
  Interventions: Procedure: Accelerated corneal collagen cross linking
- Group 2 (Epithelium-on accelerated CXL) (Active Comparator): patients with corneal thickness > 380 µm and < 400 µm thinnest location) were assigned into Epi-on Trans-epithelial accelerated CXL procedure
  Interventions: Procedure: Accelerated corneal collagen cross linking

INTERVENTIONS:
Procedure: Accelerated corneal collagen cross linking — This strategy is based on the underlying pathology of the disease. Corneal collagen cross linking (CXL) idea was based on the fact that a photosensitizer substance like riboflavin (vitamin B2) can interact with ultraviolet irradiation (Ultraviolet-A) to strengthen the corneal tissue inter and intrafibrillar collagen bonds thus preventing further thinning, corneal protrusion and reduces corneal irregular astigmatism.

SUMMARY:
Aim of work:

* To detect abnormal corneal thinning in keratoconus using pachymetry maps measured by high-speed anterior segment optical coherence tomography (OCT).
* To evaluate the visualization and depth of the demarcation line with anterior segment optical coherence tomography (AS-OCT) after corneal collagen cross-linking (CXL).
* To compare the depth of demarcation line between epithelial-on (Epi-on) and epithelial-off (Epi-off) corneal collagen cross-linking.

DETAILED DESCRIPTION:
Keratoconus is a bilateral, asymmetric, progressive, non-inflammatory corneal ectatic disorder that is characterized by progressive thinning, steepening and potential scaring. Usually it affects the inferior or central cornea that becomes thinner and bulges forward in a cone-shaped fashion, inducing irregular astigmatism and myopia and reducing the quality of vision. Approximately 50% of clinically normal fellow eyes will progress to KC within 16 years. The greatest risk is during the first 6 years of the onset.

Annual incidence of KC also varies greatly from 0.002% , to 0.23% of 100,000 population per year. Most of the western studies support the lower figure of 0.002% , while in the Middle-East it is about 0.02 per year. In the middle-East, there is about ten-fold higher incidence (0.02% compared to 0.002%), and ten-fold higher prevalence (2.34% compared to 0.23%), as compared to Western counries.

Management of keratoconus depends on a variety of factors including visual acuity, the degree of corneal thinning and steepening. Rigid gas permeable contact lenses (RGPs) have been tried to correct corneal irregularity and astigmatism in keratoconus but they don't stop keratoconus progression. Corneal collagen cross linking (CXL) is now considered as the treatment of choice in mild to moderate cases of keratoconus and is proven to halt the disease progression. The implantation of intrastromal corneal ring segments (e.g. INTACS, Ferrara & Keraring) has been indicated for cases with moderate keratoconus to flatten the steep irregular corneas. Advanced cases of keratoconus with marked deterioration of vision or corneal scarring may be good candidates for deep anterior lamellar or penetrating Keratoplasty (DALK or PKP).

Collagen cross-linking (CXL) is a relatively new conservative approach for progressive corneal ectasia, which is able to strengthen corneal tissue reforming new covalent bonds. This strategy is based on the underlying pathology of the disease. Corneal collagen cross linking (CXL) idea was based on the fact that a photosensitizer substance like riboflavin (vitamin B2) can interact with ultraviolet irradiation (Ultraviolet-A) to strengthen the corneal tissue inter and intrafibrillar collagen bonds thus preventing further thinning, corneal protrusion and reduces corneal irregular astigmatism.

Epithelial debridement enhances riboflavin corneal penetration that allows absorption of wide range of light spectrum wave lengths including ultra violet A.

The idea of trans-epithelial delivery (Epi-on technique) of riboflavin into the corneal tissue was hindered by the fact that riboflavin can't penetrate intact corneal epithelium. The addition of certain molecules such as trometamol allows penetration of riboflavin into the corneal stroma that markedly reduces the possible complications of removing of the corneal epithelium (Epi-off technique) such as persistent epithelial defects, scarring and serious infectious keratitis. Another advantage of trans-epithelial CXL that it reduces the cytotoxic effects of ultraviolet irradiation on corneal endothelium and intraocular structures especially in thin corneas less than 400 um.

Recently, CXL techniques were developed to minimize ultraviolet exposure and shorten the time of the procedure on basis of photochemical reciprocity in which increased irradiation intensity with reduced intervals achieve the same effect of the conventional cross linking techniques.

Corneal collagen cross linking induces stromal collagen fiber shrinkage. Ultraviolet A exposure enhances covalent bond formation between collagen fibers especially in the anterior stroma where 65% of ultraviolet irradiation is absorbed within first 250 um thus a hyperrefelctive transitional area can be detected between the anterior cross linked and the posterior untreated corneal stromal tissue referred to as a demarcation line that is usually evident 1 - 6 months after CXL procedure.

A comprehensive slit lamp examination could detect the demarcation line; however anterior segment ocular coherence tomography (AS-OCT) is a more sensitive tool to assess the extent and depth of a stromal demarcation line that is deeper centrally than peripherally due to the natural corneal curvature.

Several studies confirm the effectiveness and safety of conventional cross-linking procedure, which is also known as "Dresden protocol", in which the interaction between 0.1% riboflavin molecules absorbed in corneal tissue and UV-A rays delivered at 3 mW/cm2 for 30 minutes (5.4 J/cm2 energy dose) releases reactive oxygen species that promote the formation of "molecular bridges" between and within collagen fibers.

Corneal cross-linking causes a dose-dependent keratocytes damage. Wollensak et al. described cellular apoptosis to a depth of 300 µm radiating with UV- A at 3 mW/cm2. Histopathological studies showed an already complete keratocyte apoptosis limited to the anterior stroma within 24 hours. Some authors characterized the corneal stromal DL as a clinical sign to evaluate the depth of the CXL treatment.

Some studies hypothesize the role of the DL after CXL depth as representative of CXL effectiveness. Recently, the essential debate focused on whether the depth of the corneal stromal DL is indeed a true indicator of CXL efficacy. The main question is whether "the deeper, the better" principle can be applied to CXL.

In recent years, anterior segment optical coherence tomography (AS-OCT) and confocal microscopy have been used as tools to assess the depth of DL and consequently the depth of the cross-linking effect. By using the AS-OCT, the stromal DL is detected within an enhanced image of the cornea in the horizontal meridian. The image is captured when the corneal reflex is visible, and the depth of DL is measured using the caliper tool provided by the manufacturer. Doors et al described the best visibility of corneal stromal DL using AS-OCT at 1 month after CXL treatment, with an average DL depth of 313 µm; Yam et al measured the depth of DL at 6 months highlighting that the severity of ectasia and age may cause a worse DL visibility.

ELIGIBILITY:
Inclusion Criteria:

* Patients with progressive keratoconus (maximum K-reading between 46 diopters and 56 diopters), clear cornea and corneal pachymetry > 380um.

Exclusion Criteria:

* Corneal scarring.
* Advanced keratoconus (k-max > 56 D).
* Corneal pachymetry (thinnest location) < 380 µm.
* Epithelial healing disorders e.g.
* Recurrent corneal erosion syndrome.
* History of diseases that may delay corneal healing or predispose the eye for future complications (e.g. rheumatic disorders, glaucoma, uveitis, chemical burn, corneal dystrophy).
* History suggestive of herpetic keratitis because the UVR can activate herpes virus.
* Post-LASIK ectasia and/or previous corneal surgeries e.g. intrastromal corneal ring segments (INTACS).
* Pregnancy and breast-feeding.

Ages: 15 Years to 36 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 44 (Estimated)
Dates: Start 2016-10-01 (Actual); Primary Completion 2019-04 (Estimated); Study Completion 2019-05-30 (Estimated)

PRIMARY OUTCOMES:
Demarcation line (DL) depth | 3 months post corneal collagen cross linking
  DL is a hyper-reflectivity seen in the anterior corneal stroma between the crossed and non-crossed collagen stromal bundles using anterior segment optical coherence tomography.
Change in maximum keratometry (K-max) in diopters (D) | preoperative, 6 months and 12 months postoperative
  to compare preoperative values of K-max with values at both 6 and 12 months follow up visits.
Change in central corneal thickness in (µm) | preoperative, 6 months and 12 months postoperative
  using anterior segment OCT

SECONDARY OUTCOMES:
Change in visual acuity | preoperative, 6 months and 12 months postoperative
  uncorrected and best corrected visual acuity
Change in the mean refractive spherical equivalent (MRSE) | preoperative, 6 months and 12 months postoperative
  in diopters (D)
Change in pachymetry at the thinnest location | preoperative, 6 months and 12 months postoperative
  Corneal thickness at the thinnest location

CONTACTS AND LOCATIONS:
Overall Officials: Kamel Abdelnaser, MD, Study Chair — Assiut University
Locations (1):
- Teba private eye centre, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Mrochen M. Current status of accelerated corneal cross-linking. Indian J Ophthalmol. 2013 Aug;61(8):428-9. doi: 10.4103/0301-4738.116075. PMID 23925330
- [Result] Li Y, Meisler DM, Tang M, Lu AT, Thakrar V, Reiser BJ, Huang D. Keratoconus diagnosis with optical coherence tomography pachymetry mapping. Ophthalmology. 2008 Dec;115(12):2159-66. doi: 10.1016/j.ophtha.2008.08.004. Epub 2008 Nov 5. PMID 18977536
- [Result] Greenstein SA, Shah VP, Fry KL, Hersh PS. Corneal thickness changes after corneal collagen crosslinking for keratoconus and corneal ectasia: one-year results. J Cataract Refract Surg. 2011 Apr;37(4):691-700. doi: 10.1016/j.jcrs.2010.10.052. PMID 21420594